CLINICAL TRIAL: NCT05586802
Title: Dissecting the Importance of Sex Steroids Balance for Metabolic and Reproductive Health in Men With Klinefelter Syndrome: a Randomized Controlled Study
Brief Title: Sex Steroids Balance for Metabolic and Reproductive Health in Klinefelter Syndrome
Acronym: KLIN-HEALTH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Georgios Papadakis (Other)
Responsible Party: Sponsor-Investigator, Georgios Papadakis, Senior Lecturer (Privat docent & MERclin), University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PZ00P3_202151
Record Dates: First submitted 2022-10-15; First posted 2022-10-19 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Klinefelter Syndrome
Keywords: Metabolic syndrome; Infertility; Aromatase; Testosterone/estradiol ratio; mTESE biopsy; GLP1 agonists
MeSH Terms: conditions — Klinefelter Syndrome; Metabolic Syndrome; Infertility | interventions — Anastrozole; semaglutide; Chorionic Gonadotropin

STUDY DESIGN:
Intervention Model Description: Two designs according to the presence of fertility desire (Design 1) or high metabolic risk (Design 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (Fertility) - positive micro-dissection testicular sperm extraction (mTESE) biopsy 1 (No Intervention): Men with Klinefelter syndrome seeking fertility or interested in fertility preservation that undergo mTESE biopsy after wash-out of testosterone replacement therapy and have positive sperm retrieval (detectable spermatozoids)
- Group 1 (Fertility) - negative mTESE biopsy 1, then randomized to Arm A (Experimental): Men with Klinefelter syndrome seeking fertility or interested in fertility preservation that undergo mTESE biopsy after wash-out of testosterone replacement therapy and have negative sperm retrieval (no detectable spermatozoids), subsequently randomized to receive an hormonal stimulation for 26 weeks
  Interventions: Drug: Anastrozole
- Group 1 (Fertility) - negative mTESE biopsy 1, then randomized to Arm B (Experimental): Men with Klinefelter syndrome seeking fertility or interested in fertility preservation that undergo mTESE biopsy after wash-out of testosterone replacement therapy and have negative sperm retrieval (no detectable spermatozoids), subsequently randomized to receive an hormonal stimulation for 26 weeks
  Interventions: Drug: Anastrozole; Drug: human chorionic gonadotropin
- Group 2 (Metabolic Risk) - randomized to Arm C (Active Comparator): Men with Klinefelter syndrome not interested in fertility that present with high metabolic risk and consent to a wash-out of testosterone replacement therapy. They are subsequently randomized to receive an hormonal treatment to improve metabolic health. This arm will receive an active comparator by a testosterone gel
  Interventions: Drug: Testosterone gel
- Group 2 (Metabolic Risk) - randomized to Arm D (Experimental): Men with Klinefelter syndrome not interested in fertility that present with high metabolic risk and consent to a wash-out of testosterone replacement therapy. They are subsequently randomized to receive an hormonal treatment to improve metabolic health. This arm will receive an an experimental treatment
  Interventions: Drug: Anastrozole
- Group 2 (Metabolic Risk) - randomized to Arm E (Experimental): Men with Klinefelter syndrome not interested in fertility that present with high metabolic risk and consent to a wash-out of testosterone replacement therapy. They are subsequently randomized to receive an hormonal treatment to improve metabolic health. This arm will receive an an experimental treatment
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Anastrozole — This will be an experimental treatment for 26 weeks in Group 1 Arm A and Arm B as well for Group 2 Arm D
  Other Names: Anastrozole Teva
  Arms: Group 1 (Fertility) - negative mTESE biopsy 1, then randomized to Arm A; Group 1 (Fertility) - negative mTESE biopsy 1, then randomized to Arm B; Group 2 (Metabolic Risk) - randomized to Arm D
Drug: Semaglutide — This will be an experimental treatment for 26 weeks in Group 2 Arm E
  Other Names: Ozempic
  Arms: Group 2 (Metabolic Risk) - randomized to Arm E
Drug: human chorionic gonadotropin — This will be an experimental treatment for 26 weeks in addition to anastrozole in Group 1 - Arm B
  Other Names: Choriomon
  Arms: Group 1 (Fertility) - negative mTESE biopsy 1, then randomized to Arm B
Drug: Testosterone gel — This will be an active comparator for 26 weeks in Group 2 - Arm C
  Other Names: Tostran
  Arms: Group 2 (Metabolic Risk) - randomized to Arm C

SUMMARY:
The study seeks primarily to determine whether modulation of systemic and testicular sex steroids balance by aromatase inhibitors will positively affect the metabolic health and spermatogenesis of men with Klinefelter syndrome (KFS) as compared to the current state of the art for each issue.

Secondary objectives of this study are (i) to unravel the heterogeneity of the reproductive and metabolic phenotype of men with KFS by performing a multi-omic analysis in a large cohort at baseline; (ii) to evaluate the efficacy of semaglutide-induced weight loss to achieve metabolic and reproductive benefit in men with Klinefelter syndrome as compared to standard testosterone replacement; (ii) to assess whether addition of hCG to aromatase inhibitors further increases intratesticular testosterone and promotes spermatogenesis in men with KFS.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of Klinefelter syndrome (47,XXY or mosaicism)

Design 1:

* Age range: 16-40 years old
* Intention to become parent or interest in fertility preservation
* Confirmed azoospermia (lack of spermatozoids) after centrifugation of one semen sample

Design 2:

* Age range: 18-65 years old
* No interest in fertility or fertility preservation
* Hypogonadism at diagnosis or after wash-out of testosterone replacement therapy
* High metabolic risk defined as overweight (BMI 25-28 kg/m2) and insulin resistance (HOMA-IR > 2.6)

Exclusion Criteria:

* Contraindications to testosterone-rising therapies (prostate or breast cancer, PSA > 4 µg/l, active liver disease, symptomatic heart disease)
* Decreased life expectancy due to terminal disease
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study (language problems, severe psychological or mental disorders)

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Design 1 : sperm retrieval rate at mTESE biopsy | mTESE biopsy 26 weeks after hormonal intervention
  Sperm retrieval rate at mTESE biopsy (Group A and B)
Design 2 : change in insulin resistance index (HOMA-IR) | From baseline to week 26 of intervention
  HOMA-IR calculated using fasting glucose and insulin levels

CONTACTS AND LOCATIONS:
Overall Officials: GEORGIOS PAPADAKIS, MD, Principal Investigator — Service of endocrinology, diabetes & metabolism, CHUV, Lausanne University Hospital
Locations (1):
- Service of Endocrinology, Diabetes & Metabolism, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request and data transfer agreement
Supporting Information: Study Protocol, CSR
Time Frame: At study completion